CLINICAL TRIAL: NCT06080334
Title: Effectiveness of Dry Needling of the Gastrocnemius Muscle vs. Electrolysis in Subjects With Achilles Tendinopathy: a Randomised Single-blind Clinical Trial
Brief Title: Effectiveness of Dry Needling of the Gastrocnemius Muscle VS Electrolysis in Subjects With Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal investigator, Universidad Católica de Ávila
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 06/10/2023
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Achilles Tendinopathy; Pain
Keywords: achilles tendon; electrolysis; tendinopathy
MeSH Terms: conditions — Pain; Tendinopathy | interventions — Dry Needling; Electrolysis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling+eccentric exercises (Experimental): Application of dry needling on the hyperalgesic trigger points of the gastrocnemius muscle and subsequent inclusion of eccentric exercises.
  Interventions: Device: Dry needling
- Electrolysis+eccentric exercises (Experimental): Application of electrolysis to the Achilles tendon and subsequent inclusion of eccentric exercises.
  Interventions: Device: Electrolysis

INTERVENTIONS:
Device: Dry needling — Dry needling using the Hong technique on the most hyperalgesic trigger point in the gastrocnemius muscle.
  Arms: Dry needling+eccentric exercises
Device: Electrolysis — Electrolysis on the Achilles tendon using ultrasound-guided technique.
  Arms: Electrolysis+eccentric exercises

SUMMARY:
Achilles tendinopathy is the injury that primarily occurs in athletes and people who engage in repetitive activities that involve the calf muscles, such as running, jumping, and sudden acceleration and deceleration movements. To observe the effectiveness of dry needling in the PGM of the gastrocnemius muscle, in the short and medium term, on the intensity of pain in gastrocnemius muscle, in the short and medium term, on pain intensity in patients with patients with Achilles tendinopathy, compared to the application of ultrasound-guided percutaneous electrolysis on the tendon.

ELIGIBILITY:
Inclusion Criteria:

* Signing of informed consent both to participate in the study and to undergo invasive in the study, as well as to undergo invasive physiotherapy techniques. physiotherapy techniques.
* Presence of symptoms (swelling or pain) for at least 3 months.
* Positive Achilles tendon palpation test.
* Males and females over 18 years of age.
* Presence of MMP in the gastrocnemius muscle, meeting at least three of the following criteria diagnostic criteria described by Travell and Simons:
* Presence of palpable tight band.
* Local pain on pressure at the nodule of the tense band.
* Recognition by the patient as his usual pain after mechanical after mechanical stimulation of the sensitive nodule.
* Limitation of range of motion.

Exclusion Criteria:

* Any related acute or chronic musculoskeletal disease that may related chronic musculoskeletal disease, which may affect the results of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity. | 5 weeks
  Measurement of pain intensity using the VAS scale (0 minimum pain, 10 maximum bearable pain).

SECONDARY OUTCOMES:
Pressure pain threshold | 5 weeks
  Pressure pain threshold measured by algometer over the most hyperalgesic point on the Achilles tendon measured in Newtons.
Range of movement | 5 weeks
  Measurement of ankle dorsiflexion range of motion measured by digital goniometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Jorge Velázquez Saornil, Ávila, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zunko H, Vauhnik R. Reliability of the weight-bearing ankle dorsiflexion range of motion measurement using a smartphone goniometer application. PeerJ. 2021 Sep 22;9:e11977. doi: 10.7717/peerj.11977. eCollection 2021. PMID 34616594
- [Result] Kedia M, Williams M, Jain L, Barron M, Bird N, Blackwell B, Richardson DR, Ishikawa S, Murphy GA. The effects of conventional physical therapy and eccentric strengthening for insertional achilles tendinopathy. Int J Sports Phys Ther. 2014 Aug;9(4):488-97. PMID 25133077
- [Result] Lucena-Anton D, Luque-Moreno C, Valencia-Medero J, Garcia-Munoz C, Moral-Munoz JA. Effectiveness of Dry Needling of Myofascial Trigger Points in the Triceps Surae Muscles: Systematic Review. Healthcare (Basel). 2022 Sep 24;10(10):1862. doi: 10.3390/healthcare10101862. PMID 36292308
- [Result] Martin-Sacristan L, Calvo-Lobo C, Pecos-Martin D, Fernandez-Carnero J, Alonso-Perez JL. Dry needling in active or latent trigger point in patients with neck pain: a randomized clinical trial. Sci Rep. 2022 Feb 24;12(1):3188. doi: 10.1038/s41598-022-07063-0. PMID 35210467
- [Result] McDevitt AW, Snodgrass SJ, Cleland JA, Leibold MBR, Krause LA, Mintken PE. Treatment of individuals with chronic bicipital tendinopathy using dry needling, eccentric-concentric exercise and stretching; a case series. Physiother Theory Pract. 2020 Mar;36(3):397-407. doi: 10.1080/09593985.2018.1488023. Epub 2018 Jun 22. PMID 29932797
- [Result] Asensio-Olea L, Leiros-Rodriguez R, Marques-Sanchez MP, de Carvalho FO, Maciel LYS. Efficacy of percutaneous electrolysis for the treatment of tendinopathies: A systematic review and meta-analysis. Clin Rehabil. 2023 Jun;37(6):747-759. doi: 10.1177/02692155221144272. Epub 2022 Dec 30. PMID 36583575